CLINICAL TRIAL: NCT02563548
Title: A Phase 1B Open-Label Study of PEGylated Recombinant Human Hyaluronidase (PEGPH20) Combined With Pembrolizumab in Subjects With Selected Hyaluronan-High Solid Tumors
Brief Title: A Study of PEGylated Recombinant Human Hyaluronidase (PEGPH20) With Pembrolizumab in Participants With Selected Hyaluronan High Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HALO-107-101
Record Dates: First submitted 2015-08-31; First posted 2015-09-30 (Estimated); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-12

CONDITIONS: NSCLC; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — PEGPH20; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GAC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab (Experimental): Dose escalation part: Participants with relapsed/refractory locally advanced or metastatic gastric adenocarcinoma (GAC) will receive PEGPH20 1.6 micrograms/kilogram (µg/kg) or 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 milligrams/kilogram (mg/kg) every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration. Dose expansion part: Participants with relapsed/refractory locally advanced or metastatic GAC will receive PEGPH20 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle and pembrolizumab 200 mg on Day 1 of each cycle, 4-6 hours after the completion of PEGPH20 administration. Treatment in both phases of the study will continue until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 60 weeks).
  Interventions: Drug: PEGPH20; Drug: Pembrolizumab
- NSCLC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab (Experimental): Dose escalation part: Participants with relapsed/refractory Stage IIIB or IV non-small cell lung cancer (NSCLC) will receive PEGPH20 1.6 µg/kg or 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration. Dose expansion part: Participants with relapsed/refractory Stage IIIB or IV NSCLC will receive PEGPH20 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle and pembrolizumab 200 mg on Day 1 of each cycle, 4-6 hours after the completion of PEGPH20 administration. Treatment in both phases of the study will continue until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks).
  Interventions: Drug: PEGPH20; Drug: Pembrolizumab

INTERVENTIONS:
Drug: PEGPH20 — PEGPH20 will be administered as an intravenous (IV) infusion as per the dose schedule specified in the arm description.
  Other Names: PEGylated recombinant human hyaluronidase
Drug: Pembrolizumab — Pembrolizumab will be administered as an IV infusion as per the dose schedule specified in the arm description.
  Other Names: Keytruda®

SUMMARY:
This is a Phase 1b study evaluating a combination of PEGPH20 and pembrolizumab in hyaluronan-high (HA-high) participants with relapsed/refractory non-small cell lung cancer (NSCLC) and HA-high participants with relapsed/refractory gastric adenocarcinoma (GAC).

DETAILED DESCRIPTION:
Study involves dose escalation phase (completed in Nov-2016) to assess the safety and tolerability of PEGPEM (PEGylated recombinant human hyaluronidase [PEGPH20] combined with pembrolizumab [Keytruda®]) and to find the recommended Phase 2 dose (RP2D) ; and an expansion phase to assess the efficacy, safety and tolerability of PEGPEM in stage III b/IV NSCLC and relapsed/refractory GAC participants. Plan was to include approximately 51 HA-high participants (30 NSCLC and 21 GAC participants) in the dose expansion phase on the obtained RP2D from dose escalation phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Dose Expansion: Histologically confirmed and documented, previously untreated or treated stage IIIB or IV NSCLC having failed no more than 1 previous platinum containing chemotherapy regimen for locally-advanced or metastatic disease or relapsed/refractory locally advanced or metastatic gastric adenocarcinoma having failed no more than 2 previous chemotherapy regimens for locally advanced or metastatic disease. Participants with NSCLC who are known to be epidermal growth factor receptor (EGFR)-mutation positive must have received an EGFR inhibitor and participants known to be anaplastic lymphoma kinase (ALK)-mutation positive must have received an ALK inhibitor.

Prior to enrollment, confirmation of the following must be obtained:

• For participants in the dose expansion portion of the study, it is mandatory that available archived tumor tissue in formalin-fixed.

paraffin-embedded (FFPE) block or minimum 10-15 unstained consecutive core biopsy slides from 1 archival block that meet specific tissue requirements are available.

* For dose expansion: one or more tumors measurable on computed tomography (CT) scan/magnetic resonance imaging (MRI) scan per RECIST v 1.1., for dose escalation, participants need only have evaluable disease - Previously irradiated tumors may be eligible if they have clearly progressed in size.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Life expectancy greater than or equal to (≥) 3 months.

Participants must also satisfy the following inclusion criterion to be enrolled in the dose expansion portion:

* Participants (NSCLC and gastric adenocarcinoma) must be determined to have HA-high levels from their tumor biopsies.
* NSCLC and gastric adenocarcinoma participants must have tissue available for HA-selection and programmed cell death-1 (PD-L1) testing.

Exclusion Criteria:

* Previous treatment with pembrolizumab, nivolumab, or other antibody (anti-)-PD-1 or PD-1 ligand-antibody (anti-PD-L1) agents.
* New York Heart Association Class III or IV (Appendix D) cardiac disease or myocardial infarction within the past 12 months before screening, or preexisting atrial fibrillation.
* Prior history of cerebrovascular accident or transient ischemic attack.
* NSCLC participants with known brain metastases (certain exceptions allowed)
* Gastric adenocarcinoma participants with brain metastases
* History of active bleeding within the last 3 months requiring transfusion
* Anti-angiogenic therapy within the last month
* Participants with known interstitial fibrosis or interstitial lung disease.
* Previous history of pulmonary embolism or pulmonary embolism found on screening exam.
* History of:

  1. Pneumonitis that requires oral or IV steroids;
  2. Or known cases of hepatobiliary diseases (e.g., primary biliary cholangitis, primary sclerosing cholangitis, history of immune-mediated cholangitis);

     * Participants with cholangitis attributed to infectious etiology (e.g., ascending cholangitis, bacterial cholangitis) are eligible if the infection has been fully resolved prior to the screening visit.
  3. Or known cases of drug-induced hepatobiliary toxicities.
* Active autoimmune disease requiring systemic treatment within the past 3 months or documented history of clinically severe autoimmune disease, or syndrome that requires systemic steroids or immunosuppressive agents.
* History of another primary cancer within the last 3 years that required treatment, with the exception of non-melanoma skin cancer, early-stage prostate cancer, or curatively treated cervical carcinoma in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Development, Study Director — Halozyme Therapeutics
Locations (28):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona, Scottsdale, Arizona
  - California Cancer Associates for Research and Excellence - Encinitas, Encinitas, California
  - University of California San Diego - Moores Cancer Center, La Jolla, California
  - St. Joseph's Hospital, Orange, California
  - University of California - Davis, Sacramento, California
  - St. Joseph's Hospital, Santa Rosa, California
  - Innovative Clinical Research, Whittier, California
  - University of Colorado Denver University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Holy Cross Hospitals, Fort Lauderdale, Florida
  - University of Miami/Sylvester Cancer Center, Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - New Jersey Hematology Oncology Associates, Brick, New Jersey
  - University of Rochester, Rochester, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Swedish Health Services, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts: dose escalation and dose expansion. A total of 56 participants were enrolled (35 with gastric adenocarcinoma [GAC] and 21 with non-small cell lung cancer [NSCLC]).
Pre-assignment Details: 14 participants (10 with GAC and 4 with NSCLC) were enrolled in dose escalation part. Due to evolving standard-of-care in the immuno-oncology treatment landscape, this study discontinued further enrollment on 31 May 2018. At the time of the early termination, 42 participants (25 with GAC and 17 with NSCLC) had been enrolled in dose expansion part.
Groups:
- Dose Escalation (GAC): PEGPH20 1.6 µg/kg + Pembrolizumab: Participants with relapsed/refractory locally advanced or metastatic GAC received PEGylated recombinant human hyaluronidase (PEGPH20) 1.6 micrograms/kilogram (µg/kg) on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 milligrams/kilogram (mg/kg) every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks).
- Dose Escalation (NSCLC): PEGPH20 1.6 µg/kg + Pembrolizumab: Participants with relapsed/refractory Stage IIIB or IV NSCLC received PEGPH20 1.6 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 27 weeks).
- Dose Escalation (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab: Participants with relapsed/refractory locally advanced or metastatic GAC received PEGPH20 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks).
- Dose Escalation (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab: Participants with relapsed/refractory Stage IIIB or IV NSCLC received PEGPH20 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 27 weeks).
- Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab: Participants with relapsed/refractory locally advanced or metastatic GAC received PEGPH20 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle and pembrolizumab 200 mg on Day 1 of each cycle, 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 60 weeks).
- Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab: Participants with relapsed/refractory Stage IIIB or IV NSCLC received PEGPH20 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle and pembrolizumab 200 mg on Day 1 of each cycle, 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks).
Period: Dose Escalation (Up to 46 Weeks)
Arm/Group | Dose Escalation (GAC): PEGPH20 1.6 µg/kg + Pembrolizumab | Dose Escalation (NSCLC): PEGPH20 1.6 µg/kg + Pembrolizumab | Dose Escalation (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Escalation (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Started | 3 | 2 | 7 | 2 | 0 | 0
Received at Least 1 Dose of Study Drug | 3 | 2 | 7 | 2 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 7 | 2 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Radiological Progression | 1 | 2 | 2 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 0 | 0
Period: Dose Expansion (Up to 60 Weeks)
Arm/Group | Dose Escalation (GAC): PEGPH20 1.6 µg/kg + Pembrolizumab | Dose Escalation (NSCLC): PEGPH20 1.6 µg/kg + Pembrolizumab | Dose Escalation (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Escalation (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Started | 0 | 0 | 0 | 0 | 25 | 17
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 24 | 17
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 25 | 17
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 8
Not completed — Radiological Progression | 0 | 0 | 0 | 0 | 15 | 3
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 6 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Investigator or Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Increased brain lesions | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Enrolled but not treated | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included participants who received at least 1 dose of any study medication (PEGPH20 or pembrolizumab) in either dose escalation or dose expansion portion of the study.
Groups:
- GAC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab: Dose escalation part: Participants with relapsed/refractory locally advanced or metastatic GAC received PEGPH20 1.6 µg/kg or 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration.
  Dose expansion part: Participants with relapsed/refractory locally advanced or metastatic GAC received PEGPH20 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle and pembrolizumab 200 mg on Day 1 of each cycle, 4-6 hours after the completion of PEGPH20 administration.
  Treatment in both phases of the study was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 60 weeks).
- NSCLC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab: Dose escalation part: Participants with relapsed/refractory Stage IIIB or IV NSCLC received PEGPH20 1.6 µg/kg or 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration.
  Dose expansion part: Participants with relapsed/refractory Stage IIIB or IV NSCLC received PEGPH20 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle and pembrolizumab 200 mg on Day 1 of each cycle, 4-6 hours after the completion of PEGPH20 administration.
  Treatment in both phases of the study was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks).
- Total: Total of all reporting groups
Arm/Group | GAC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab | NSCLC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab | Total
Number analyzed (Participants) | 34 | 21 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.89) | 67.7 (10.66) | 64.4 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 29 | 10 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 32 | 18 | 50
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 30 | 17 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose-Escalation Phase: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: DLTs were defined as any of the following: i) Any treatment-emergent Grade greater than or equal to (≥) 3 toxicity that was considered related to either PEGPH20 or pembrolizumab or the combination of PEGPH20 and pembrolizumab (nausea, vomiting, MSEs, and diarrhea were considered DLTs only if they reached Grade ≥ 3 despite adequate supportive care measures); ii) Grade 3 musculoskeletal events (MSEs) were considered DLTs only if they did not reduce to Grade ≤ 2 within 48 hours despite therapeutic intervention; iii) Hypersensitivity/infusion reactions related to PEGPH20 or pembrolizumab dosing were not considered DLTs (hypersensitivity reactions were generally not related to the dose level of a drug since they could occur even upon a low level of exposure).
Time Frame: Cycle 1 (21 days)
Population: DLT evaluable population included all participants enrolled in dose escalation part who received at least 1 of the 3 full planned doses of PEGPH20 and 1 complete dose of pembrolizumab in Cycle 1 and had been followed for the first 21 days of treatment or had experienced a DLT during the initial 21 days (Cycle 1) of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation (GAC): PEGPH20 1.6 µg/kg + Pembrolizumab: Participants with relapsed/refractory locally advanced or metastatic GAC received PEGPH20 1.6 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks).
Arm/Group | Dose Escalation (GAC): PEGPH20 1.6 µg/kg + Pembrolizumab | Dose Escalation (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Escalation (NSCLC): PEGPH20 1.6 µg/kg + Pembrolizumab | Dose Escalation (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 2 | 7 | 2 | 2
Participants | 0 | 0 | 0 | 1

2. Primary Outcome: Dose-Escalation Phase: Maximum Tolerated Dose (MTD) of PEGPH20 in Combination With Pembrolizumab
Description: MTD of PEGPEM combination (PEGPH20 + Pembrolizumab) was defined as the highest dose level at which no more than 1 of 6 evaluable participants had experienced a DLT in the first 3 weeks of treatment. DLT was defined as any of the following: i) Any treatment-emergent Grade greater than or equal to (≥) 3 toxicity that was considered related to either PEGPH20 or pembrolizumab or the combination of PEGPH20 and pembrolizumab (nausea, vomiting, MSEs, and diarrhea were considered DLTs only if they reached Grade ≥ 3 despite adequate supportive care measures); ii) Grade 3 musculoskeletal events (MSEs) were considered DLTs only if they did not reduce to Grade ≤ 2 within 48 hours despite therapeutic intervention; iii) Hypersensitivity/infusion reactions related to PEGPH20 or pembrolizumab dosing were not considered DLTs (hypersensitivity reactions were generally not related to the dose level of a drug since they could occur even upon a low level of exposure).
Time Frame: Cycle 1 (21 days)
Population: After 9 participants enrolled in "Dose Escalation: PEGPH20 2.2 µg/kg + Pembrolizumab" group with only 1 DLT, the Sponsor decided to stop further dose escalation beyond 2.2 μg/kg, hence MTD was not established.
Arm/Group | Dose Escalation (GAC): PEGPH20 1.6 µg/kg + Pembrolizumab | Dose Escalation (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Escalation (NSCLC): PEGPH20 1.6 µg/kg + Pembrolizumab | Dose Escalation (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Dose Escalation Phase: Recommended Phase 2 Dose (RP2D) of PEGPH20 in Combination With Pembrolizumab
Description: The RP2D was determined based on the overall safety profile of the participants enrolled during the dose-escalation part of the study.
Time Frame: Cycle 1 (21 days)
Population: as for outcome 1
Measure: Number; unit: µg/kg
Groups:
- Dose Escalation Phase: All Participants (GAC and NSCLC): Participants with relapsed/refractory locally advanced or metastatic GAC or Stage IIIB or IV NSCLC received PEGPH20 1.6 µg/kg or 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks for GAC, and 27 weeks for NSCLC).
Arm/Group | Dose Escalation Phase: All Participants (GAC and NSCLC)
Number analyzed (Participants) | 13
µg/kg | 2.2

4. Primary Outcome: Dose Expansion Phase: Objective Response Rate (ORR): Percentage of Participants With Objective Response, as Assessed by Investigator Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: ORR was defined as percentage of participants who achieved either a complete response (CR) or partial response (PR), as assessed by investigator based on RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions; Any pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Cycle 1 Day 1 of dose-expansion phase until death, disease progression, or unacceptable toxicity (maximum exposure: 60 weeks for GAC, and 46 weeks for NSCLC)
Population: Tumor response evaluable population included all hyaluronan- high (HA-high) participants who received at least 1 dose of the RP2D of PEGPH20 and at least 1 dose of pembrolizumab; and who had at least one post-baseline tumor assessment on or post Cycle 2.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 21 | 14
percentage of participants | 9.5 [2.6 to 23.4] | 28.6 [13.1 to 49.2]

5. Secondary Outcome: Dose-Escalation Phase: ORR: Percentage of Participants With Objective Response, as Assessed by Investigator Based on RECIST Version 1.1
Description: ORR was defined as percentage of participants who achieved either a CR or PR, as assessed by investigator based on RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions; Any pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Cycle 1 Day 1 of dose-escalation phase until death, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks for GAC, and 27 weeks for NSCLC)
Population: Tumor response evaluable population included all HA-high participants who received at least 1 dose of the RP2D of PEGPH20 and at least 1 dose of pembrolizumab; and who had at least one post-baseline tumor assessment on or post Cycle 2.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Dose Escalation (GAC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab: Participants with relapsed/refractory locally advanced or metastatic GAC received PEGPH20 1.6 µg/kg or 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks).
- Dose Escalation(NSCLC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab: Participants with relapsed/refractory Stage IIIB or IV NSCLC received PEGPH20 1.6 µg/kg or 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 27 weeks).
Arm/Group | Dose Escalation (GAC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab | Dose Escalation(NSCLC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab
Number analyzed (Participants) | 8 | 3
percentage of participants | 0 [0.0 to 25.0] | 0 [0.0 to 53.6]

6. Secondary Outcome: Dose-Escalation and Expansion Phase: Duration of Response (DOR), as Assessed by Investigator Based on RECIST v1.1
Description: DOR was defined as the time from the date on which objective response (CR or PR) was first determined until the first date on which radiographic disease progression was determined. CR was defined as disappearance of all target and non-target lesions; Any pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study thus far, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of one or more new lesions; and unequivocal progression of existing non-target lesions. DOR was analyzed using Kaplan-Meier methods.
Time Frame: From date of first objective response (CR or PR) until date of first radiographic disease progression (maximum exposure: 46 weeks for GAC, and 27 weeks for NSCLC in dose-escalation; 60 weeks for GAC, and 46 weeks for NSCLC in dose-expansion)
Population: Tumor response evaluable population included all HA-high participants who received at least 1 dose of the RP2D of PEGPH20 and at least 1 dose of pembrolizumab; and who had at least one post-baseline tumor assessment on or post Cycle 2. 'Overall number of participants analyzed'=participants with a confirmed objective response.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Dose Escalation (GAC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab | Dose Escalation(NSCLC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 0 | 0 | 2 | 4
months |  |  | 8.5 [NA to NA] — Due to less number of participants with an event, upper and lower limit of 80% CI could not be calculated. | 2.8 [1.3 to 2.8]

7. Secondary Outcome: Dose-Escalation and Expansion Phase: Disease Control Rate (DCR), as Assessed by Investigator Based on RECIST v1.1: Percentage of Participants Who Achieved CR, PR or Stable Disease (SD)
Description: DCR was defined as percentage of participants who achieved CR, PR, or stable disease (SD). CR was defined as disappearance of all target and non-target lesions; Any pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study thus far, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of one or more new lesions; and unequivocal progression of existing non-target lesions.
Time Frame: From first dose until first occurrence of CR, PR or SD (maximum exposure: 46 weeks for GAC, and 27 weeks for NSCLC in dose-escalation phase; maximum exposure: 60 weeks for GAC, and 46 weeks for NSCLC in dose-expansion phase)
Population: as for outcome 5
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation (GAC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab | Dose Escalation(NSCLC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 8 | 3 | 21 | 14
percentage of participants | 12.5 [1.3 to 40.6] | 66.7 [19.6 to 96.5] | 47.6 [32.1 to 63.6] | 71.4 [50.8 to 86.9]

8. Secondary Outcome: Dose-Escalation and Expansion Phase: Progression-Free Survival (PFS), as Assessed by Investigator Based on RECIST v1.1
Description: PFS was defined as the time from first dose date until the first occurrence of either radiographic or clinical disease progression as determined by the Investigator or death from any cause before discontinuation from treatment. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study thus far, the sum must also demonstrate an absolute increase of at least 5 mm, or the appearance of one or more new lesions; and unequivocal progression of existing non-target lesions. PFS was analyzed using Kaplan-Meier methods.
Time Frame: From first dose until first occurrence of either radiographic or clinical disease progression or death (maximum exposure: 46 weeks for GAC, and 27 weeks for NSCLC in dose-escalation; 60 weeks for GAC, and 46 weeks for NSCLC in dose-expansion)
Population: Efficacy evaluable population included all HA-high participants who received at least 1 dose of the RP2D of PEGPH20 and at least 1 dose of pembrolizumab.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Dose Escalation (GAC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab | Dose Escalation(NSCLC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 10 | 4 | 24 | 17
months | 1.2 [1.2 to 1.4] | 1.7 [0.9 to NA] — Due to less number of participants with an event, upper limit of 80% CI could not be calculated. | 1.4 [1.2 to 1.4] | 4.2 [1.7 to 5.8]

9. Secondary Outcome: Dose-Escalation and Expansion Phase: Overall Survival
Description: Overall survival was defined as the time from first dose date until death from any cause. Overall survival was analyzed using Kaplan-Meier methods.
Time Frame: From first dose until death from any cause (maximum exposure: 46 weeks for GAC, and 27 weeks for NSCLC in dose-escalation phase; maximum exposure: 60 weeks for GAC, and 46 weeks for NSCLC in dose-expansion phase)
Population: as for outcome 8
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Dose Escalation (GAC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab | Dose Escalation(NSCLC): PEGPH20 1.6 or 2.2 µg/kg+Pembrolizumab | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 10 | 4 | 24 | 17
months | 2.9 [1.8 to 7.5] | 4.7 [2.8 to NA] — Due to fewer number of participants with an event, upper limit of 80% CI could not be calculated. | 4.4 [3.5 to 5.8] | 12.9 [5.1 to NA] — Due to fewer number of participants with an event, upper limit of 80% CI could not be calculated.

10. Secondary Outcome: Dose Expansion Phase: Objective Response Rate (ORR): Percentage of Participants With Objective Response, as Assessed by Investigator Based on Immune-Response Related Criteria (irRC)
Description: ORR was defined as percentage of participants who achieved either CR or PR, as assessed by investigator based on irRC. CR was defined as disappearance of all lesions including non-index lesions and new non-measurable lesions, lymph nodes must be <10 mm in short axis). PR was defined as at least a 30% decrease in tumor burden from baseline.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 21 | 14
percentage of participants | 9.5 [2.6 to 23.4] | 28.6 [13.1 to 49.2]

11. Secondary Outcome: Dose- Expansion Phase: DOR, as Assessed by Investigator Based on irRC
Description: DOR was defined as the time from the date on which objective response (CR or PR) was first determined until the first date on which radiographic disease progression was determined. CR was defined as disappearance of all lesions including non-index lesions and new non-measurable lesions, lymph nodes must be <10 mm in short axis). PR was defined as at least a 30% decrease in tumor burden from baseline. Disease progression was defined as at least a 20% increase in tumor burden from nadir. DOR was analyzed using Kaplan-Meier methods.
Time Frame: From the date of first objective response (CR or PR) until the date of first radiographic disease progression (maximum exposure: 60 weeks for GAC, and 46 weeks for NSCLC)
Population: as for outcome 6
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 2 | 4
months | 8.5 [NA to NA] — Due to fewer number of participants with an event, upper and lower limit of 80% CI could not be calculated. | 2.8 [1.3 to 2.8]

12. Secondary Outcome: Dose- Expansion Phase: DCR, as Assessed by Investigator Based on irRC: Percentage of Participants Who Achieved CR, PR or SD
Description: DCR was defined as percentage of participants who achieved CR, PR, or stable disease (SD). CR was defined as disappearance of all lesions including non-index lesions and new non-measurable lesions, lymph nodes must be <10 mm in short axis). PR was defined as at least a 30% decrease in tumor burden from baseline. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in tumor burden from nadir.
Time Frame: From first dose until first occurrence of CR, PR or SD (maximum exposure: 60 weeks for GAC, and 46 weeks for NSCLC)
Population: as for outcome 5
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 21 | 14
percentage of participants | 47.6 [32.1 to 63.6] | 78.6 [58.3 to 91.9]

13. Secondary Outcome: Dose- Expansion Phase: PFS, as Assessed by Investigator Based on irRC
Description: PFS was defined as the time from first dose date until the first occurrence of either radiographic or clinical disease progression as determined by the Investigator or death from any cause before discontinuation from treatment. Disease progression was defined as at least a 20% increase in tumor burden from nadir. PFS was analyzed using Kaplan-Meier methods.
Time Frame: From first dose until the first occurrence of either radiographic or clinical disease progression or death from any cause (maximum exposure: 60 weeks for GAC, and 46 weeks for NSCLC)
Population: as for outcome 8
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Dose Expansion (GAC): PEGPH20 2.2 µg/kg + Pembrolizumab | Dose Expansion (NSCLC): PEGPH20 2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 24 | 17
months | 1.4 [1.2 to 1.4] | 4.2 [1.7 to 5.8]

14. Secondary Outcome: Dose-Escalation and Expansion Phase: Maximum Observed Plasma Concentration (Cmax) of PEGPH20
Description: Pharmacokinetic (PK) parameters for PEGPH20 were calculated using noncompartmental methods and summarized using descriptive statistics by dose.
Time Frame: Pre PEGPH20 dose (within 2 hours [hrs] pre-dose); 0.25,1, 2-4, and 6-8 hrs post PEGPH20 dose at Cycle 1 Day 1 (cycle length = 21 days)
Population: Evaluable PK population included participants with at least one PK parameter for PEGPH20 following dosing on Day 1 of Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- PEGPH20 1.6 μg/kg + Pembrolizumab 2 mg/kg: Participants with relapsed/refractory locally advanced or metastatic GAC or relapsed/refractory Stage IIIB or IV NSCLC received PEGPH20 1.6 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration in dose escalation phase of study. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks in participants with GAC and 27 weeks in participants with NSCLC).
- PEGPH20 2.2 μg/kg + Pembrolizumab 2 mg/kg: Participants with relapsed/refractory locally advanced or metastatic GAC or relapsed/refractory Stage IIIB or IV NSCLC received PEGPH20 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle (i.e. 3 doses/cycle) and pembrolizumab 2 mg/kg every 21 days on Day 1 of each cycle (i.e. 1 dose/cycle), 4-6 hours after the completion of PEGPH20 administration in dose escalation phase of study. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 46 weeks in participants with GAC and 27 weeks in participants with NSCLC).
- PEGPH20 2.2 μg/kg + Pembrolizumab 200 mg: Participants with relapsed/refractory locally advanced or metastatic GAC or relapsed/refractory Stage IIIB or IV NSCLC received PEGPH20 2.2 µg/kg on Day 1, Day 8 and Day 15 of each 21-day cycle and pembrolizumab 200 mg on Day 1 of each cycle, 4-6 hours after the completion of PEGPH20 administration. Treatment was continued until death, withdrawal of consent from the study, disease progression, or unacceptable toxicity (maximum exposure: 60 weeks in participants with GAC and 46 weeks in participants with NSCLC).
Arm/Group | PEGPH20 1.6 μg/kg + Pembrolizumab 2 mg/kg | PEGPH20 2.2 μg/kg + Pembrolizumab 2 mg/kg | PEGPH20 2.2 μg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 8 | 40
nanograms/milliliter (ng/mL) | 38.3 (21.4) | 48.7 (26.4) | 54.1 (21.7)

15. Secondary Outcome: Dose-Escalation and Expansion Phase: Terminal Elimination Half-Life (t1/2) of PEGPH20
Description: PK parameters for PEGPH20 were calculated using noncompartmental methods and summarized using descriptive statistics by dose.
Time Frame: as for outcome 14
Population: Evaluable PK population included participants with at least one PK parameter for PEGPH20 following dosing on Day 1 of Cycle 1. 'Overall number of participants analyzed'=participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PEGPH20 1.6 μg/kg + Pembrolizumab 2 mg/kg | PEGPH20 2.2 μg/kg + Pembrolizumab 2 mg/kg | PEGPH20 2.2 μg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 4 | 7 | 37
hours | 23.7 (5.25) | 21.8 (8.98) | 24.9 (5.76)

16. Secondary Outcome: Dose-Escalation and Expansion Phase: Area Under the Plasma Concentration Vs. Time Curve From Time 0 to Last Quantifiable Concentration (AUClast) of PEGPH20
Description: as for outcome 15
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | PEGPH20 1.6 μg/kg + Pembrolizumab 2 mg/kg | PEGPH20 2.2 μg/kg + Pembrolizumab 2 mg/kg | PEGPH20 2.2 μg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 8 | 40
h*ng/mL | 579 (18.3) | 698 (48.7) | 822 (31.9)

17. Secondary Outcome: Dose-Escalation and Expansion Phase: Volume of Distribution (Vd) of PEGPH20
Description: as for outcome 15
Time Frame: as for outcome 14
Population: Vd could not be determined due to the AUC% extrapolation of greater than 20%.
Arm/Group | PEGPH20 1.6 μg/kg + Pembrolizumab 2 mg/kg | PEGPH20 2.2 μg/kg + Pembrolizumab 2 mg/kg | PEGPH20 2.2 μg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Dose-Escalation and Expansion Phase: Clearance (CL) of PEGPH20
Description: as for outcome 15
Time Frame: as for outcome 14
Population: CL could not be determined due to the AUC% extrapolation of greater than 20%.
Arm/Group | PEGPH20 1.6 μg/kg + Pembrolizumab 2 mg/kg | PEGPH20 2.2 μg/kg + Pembrolizumab 2 mg/kg | PEGPH20 2.2 μg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Cycle 1 Day 1 up to 30 days after last dose of study drug (maximum exposure: 60 weeks for GAC, and 46 weeks for NSCLC)
Population: Safety population included all enrolled participants in either the Dose Escalation or Dose Expansion portion of the study, who received at least 1 dose of any study medication (PEGPH20 or pembrolizumab).
Measure: Count of Participants; unit: Participants
Arm/Group | GAC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab | NSCLC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 34 | 21
Participants | 34 | 21

20. Secondary Outcome: Dose-Expansion Phase: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Parameters and Vital Signs
Description: Clinical laboratory parameters included hematology (haemoglobin [Hb], hematocrit, red blood cell count, white blood cell count, neutrophils [ANC], lymphocytes, monocytes, eosinophils, basophils, granulocytes, mean corpuscular Hb, mean corpuscular volume, and platelet count) and blood chemistry (glucose, blood urea nitrogen [BUN], alanine aminotransferase [ALT], aspartate aminotransferase [AST], albumin, bilirubin, bicarbonate, calcium, chloride, magnesium, potassium, sodium, thyrotropin, thyroxin, triiodothyronine, alkaline phosphatase [ALP], electrolytes, and creatinine). Vital signs included measurement of blood pressure (systolic and diastolic), pulse, respiratory rate, and body temperature. Criteria for clinical significance were as per investigator's discretion.
Time Frame: Cycle 1 Day 1 up to 30 days after last dose of study drug (maximum exposure: 60 weeks for GAC, and 46 weeks for NSCLC)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GAC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab | NSCLC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 34 | 21
Participants | 0 | 0

21. Secondary Outcome: Dose-Expansion Phase: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG)
Description: ECGs including clinical significance was evaluated by the Investigator. Criteria for clinical significance were as per investigator's discretion.
Time Frame: Cycle 1 Day 1 up to 30 days after last dose of study drug (maximum exposure: 60 weeks for GAC, and 46 weeks for NSCLC)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GAC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab | NSCLC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab
Number analyzed (Participants) | 34 | 21
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Cycle 1 Day 1 up to 30 days after last dose of study drug (maximum exposure: 60 weeks for GAC, and 46 weeks for NSCLC)
Description: Safety population included all enrolled participants in either the Dose Escalation or Dose Expansion portion of the study, who received at least 1 dose of any study medication (PEGPH20 or pembrolizumab). Safety data was collected and summarized by cancer type (i.e., GAC and NSCLC).
Arm/Group | GAC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab | NSCLC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/34 | 2/21
Serious Adverse Events (participants affected / at risk) | 10/34 | 8/21
Other Adverse Events (participants affected / at risk) | 33/34 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GAC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab (N=34) | NSCLC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab (N=21)
Pneumonia (Infections and infestations) | 1 | 4
Sepsis (Infections and infestations) | 0 | 1
Stoma site infection (Infections and infestations) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GAC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab (N=34) | NSCLC: PEGPH20 1.6 µg/kg/2.2 µg/kg + Pembrolizumab (N=21)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 12 | 8
Vomiting (Gastrointestinal disorders) | 9 | 5
Abdominal pain (Gastrointestinal disorders) | 8 | 5
Constipation (Gastrointestinal disorders) | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Abdominal distension (Gastrointestinal disorders) | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 0
Oedema peripheral (General disorders) | 13 | 6
Fatigue (General disorders) | 12 | 6
Asthenia (General disorders) | 3 | 1
Pyrexia (General disorders) | 3 | 1
Peripheral swelling (General disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 8 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 3 | 0
Weight decreased (Investigations) | 5 | 3
Blood creatinine increased (Investigations) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
Due to evolving standard-of-care in the immuno-oncology treatment landscape, this study discontinued further enrollment on 31 May 2018.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT02563548/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT02563548/SAP_001.pdf